CLINICAL TRIAL: NCT04397289
Title: The Preventive Effect of Anticoagulants on the Formation of Thrombosis After Splenectomy in Liver Cirrhosis Patients With Portal Hypertension
Brief Title: Anticoagulation Therapy After Splenectomy in Cirrhosis Patient
Acronym: ATASICP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: XJTU1AF2017LSK-43
Record Dates: First submitted 2019-11-06; First posted 2020-05-21 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Liver Cirrhosis; Portal Hypertension; Anticoagulant-induced Bleeding; Thrombosis
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Thrombosis | interventions — Heparin; Rivaroxaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Heparin group (Experimental): Low molecular weight heparin 5000U ih Q12h was given 24 hours after operation, 5 days after operation. Warfarin 1.25-2.5 mg po qd, 30 days after operation. PT/INR was kept at 1.25-1.5.
  Interventions: Drug: Heparin and Rivaroxaban
- Rivaroxaban group (Experimental): Rivaroxaban 10mg PO QD from 24 hours after operation, 30 days after operation. PT/INR was kept at 1.25-1.5.
  Interventions: Drug: Heparin and Rivaroxaban
- Control group (Sham Comparator): No preventive intervention measures.
  Interventions: Drug: Heparin and Rivaroxaban

INTERVENTIONS:
Drug: Heparin and Rivaroxaban — Low molecular weight heparin 5000U ih Q12h was given 24 hours after operation, 5 days after operation Rivaroxaban 10mg PO QD from 24 hours after operation, 30 days after operation
  Other Names: platelet collection

SUMMARY:
1. Inclusion and Exclusion Criteria Inclusion criteria: Inpatients who received laparotomy or laparoscopic splenectomy according to clinical, B-ultrasound scan, CT or MRI diagnosis of cirrhosis and portal hypertension.

Exclusion criteria:

1. ) Portal vein system thrombosis (PVST) found by preoperative color Doppler ultrasound or MRI examination;
2. ) Liver cirrhosis complicated with liver tumor;
3. ) Liver cirrhosis complicated with blood system diseases;
4. ) Patients who have not signed the informed consent form.

2. Research subgroup According to the order of the patients, the following groups are entered in turn, and the cycle is repeated.

1. ) Heparin group
2. ) Rivaroxaban group
3. ) Control group.

DETAILED DESCRIPTION:
1. Inclusion and Exclusion Criteria Inclusion criteria: Inpatients who received laparotomy or laparoscopic splenectomy according to clinical, B-ultrasound scan, CT or MRI diagnosis of cirrhosis and portal hypertension.

Exclusion criteria:

1. ) Portal vein system thrombosis (PVST) found by preoperative color Doppler ultrasound or MRI examination;
2. ) Liver cirrhosis complicated with liver tumor;
3. ) Liver cirrhosis complicated with blood system diseases;
4. ) Patients who have not signed the informed consent form.

2. Research subgroup According to the order of the patients, the following groups are entered in turn, and the cycle is repeated.

1. ) Heparin group: Low molecular weight heparin 5000U ih Q12h was given 24 hours after operation, 5 days after operation. Warfarin 1.25-2.5 mg po qd, 30 days after operation. PT（prothrombin time）/INR（international normalized ratio） was kept at 1.25-1.5.
2. ) Rivaroxaban group: Rivaroxaban 10mg po qd from 24 hours after operation, 30 days after operation. PT/INR was kept at 1.25-1.5.
3. ) Control group: No preventive intervention measures. If platelets in the above groups are > 500× 109/L, aspirin 100 mg qd is added for 1 month. If platelets are > 1000× 109/L, platelet collection is performed.

3. Monitoring indicators Color Doppler ultrasound was reexamined 1, 2, 3 and 4 weeks after operation to find out whether PVST was present. Abdominal CT was performed when PVST was suspected. After the patient's condition is stable, the portal vein system ultrasound is reviewed monthly, and the follow-up time is 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients who received laparotomy or laparoscopic splenectomy according to clinical, B-ultrasound scan, CT or MRI diagnosis of cirrhosis and portal hypertension

Exclusion Criteria:

* Portal vein thrombosis found by preoperative color Doppler ultrasound or MRI examination;
* Liver cirrhosis complicated with liver tumor;
* Liver cirrhosis complicated with blood system diseases;
* Patients who have not signed the informed consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
thrombosis formation | 1 year after surgery.
  The evaluation index is the incidence of PVST

CONTACTS AND LOCATIONS:
Overall Officials: yingmin yao, PhD, Study Director — the first hospital of xi'an jiaotong university
Locations (1):
- the first hospital of xi'an jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No